CLINICAL TRIAL: NCT03216928
Title: Pilot Study Investigating a New Mode of Action of Anti-TNF, Reverse Signaling, in Rheumatoid Arthritis
Brief Title: A New Mode of Action of Anti-TNF, Reverse Signaling, in Rheumatoid Arthritis
Acronym: TNF-RS-PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15 7735 02
Record Dates: First submitted 2017-06-12; First posted 2017-07-13 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Reverse Signaling; Anti-TNF
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): patients with good response to anti-TNF had a blood test
  Interventions: Diagnostic Test: Blood test
- Group 2 (Experimental): patients with moderate or non-response to anti-TNF had a blood test
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test

SUMMARY:
Blood test in Rheumatoid Arthritis (RA) patients with good response to anti-Tumor Necrosis Factor (anti-TNF) and in patients with moderate or non-response will be done in the month following the evaluation of clinical response to therapy. Isolation of mononuclear cells and purification of monocyte by negative selection. Cell culture of monocyte in presence or not of anti-TNF for 24 hours and analyze of CD36 (cluster of differentiation antigen 36) expression (principal outcome). For secondary outcomes analyze monocyte phenotype, NRF2 nuclear translocation, and clinical data of patients.

ELIGIBILITY:
Inclusion Criteria:

* RA defined according to the American College of Rheumatology (ACR) 2010 criteria,
* treated by anti-TNF + methotrexate, good responders in in one arm, and moderate or non-responders in the other arm according to EULAR (European Ligue Against Rheumatism) response criteria after three months of treatment

Exclusion Criteria:

* contra-indication to anti-TNF
* corticosteroid more than 10mg by a day equivalent prednisone,
* modification of DMARD (disease-modifying antirheumatic drugs) in the last three months
* comprehension trouble
* Factors modifying CD36 -cluster of differentiation antigen 36- expression as diabetes mellitus, kidney disease, HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
CD36 expression | Day 0
  Percentage of increase of CD36 (cluster of differentiation 36) expression induced by anti-TNF ex vivo after 24h of cell culture in two groups of human monocytes: monocytes providing of RA patients good responder to anti-TNF in one hand, and moderate or non-responder in the other hand.

SECONDARY OUTCOMES:
Monocytes | Day 0
  Phenotype of freshly isolated monocytes before cell-culture
Nuclear translocation of NRF2 | Day 0
  Nuclear translocation of Nuclear factor (erythroid-derived 2)-like 2 (NRF2) induced by anti-TNF ex vivo

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Frédéric Boyer, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No